CLINICAL TRIAL: NCT07285473
Title: Low-dose Naltrexone (LDN) for the Treatment of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS): Dose-Finding
Brief Title: Low-Dose Naltrexone For ME/CFS: Dose-Finding
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jarred Younger, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300015917; 1UG3NS141843 (Other: NINDS)
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Keywords: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome; ME/CFS
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Naltrexone

STUDY DESIGN:
Masking Description: This study is single-blind, participants will not know when they received 1.5mg/day, 3.0mg/day, 4.5mg/day, or 6.0mg/day low-dose naltrexone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants Receiving Low-Dose Naltrexone (Experimental): Participants Receiving Low-Dose Naltrexone
  Interventions: Drug: Low-Dose Naltrexone, 1.5mg; Drug: Low-Dose Naltrexone, 3.0mg; Drug: Low-Dose Naltrexone, 4.5mg; Drug: Low-Dose Naltrexone, 6.0mg

INTERVENTIONS:
Drug: Low-Dose Naltrexone, 1.5mg — Low-Dose Naltrexone (LDN) is not a commercially available drug and will be compounded for this study. LDN will be taken orally, up to once per day.
  Other Names: Naltrexone
Drug: Low-Dose Naltrexone, 3.0mg — Low-Dose Naltrexone (LDN) is not a commercially available drug and will be compounded for this study. LDN will be taken orally, up to once per day.
  Other Names: Naltrexone
Drug: Low-Dose Naltrexone, 4.5mg — Low-Dose Naltrexone (LDN) is not a commercially available drug and will be compounded for this study. LDN will be taken orally, up to once per day.
  Other Names: Naltrexone
Drug: Low-Dose Naltrexone, 6.0mg — Low-Dose Naltrexone (LDN) is not a commercially available drug and will be compounded for this study. LDN will be taken orally, up to once per day.
  Other Names: Naltrexone

SUMMARY:
This exploratory clinical trial tests low-dose naltrexone (LDN) for the treatment of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS). A remote trial approach is used, with eligibility open to the state of Alabama.

DETAILED DESCRIPTION:
This study uses a remote design where individuals can participate from anywhere in the state of Alabama. Study medications will be received by mail. All participants must meet ME-ICC criteria. This study will be tested on participants recruited nationwide, with a total of 75 participants enrolled for the entire study. Participation will last 10 months.

The first stage of the study is the baseline phase. During this time, participants will complete weekly outcome measurements but will not take any medications. The baseline stage will last for 30 days. This period is used to calculate a stable baseline for determining treatment effects. After the 30-day baseline, the treatment stage will begin.

After the baseline period, participants will receive LDN capsules at one of four doses: 1.5mg/day, 3.0mg/day, 4.5mg/day, and 6.0mg/day in a blinded fashion. Capsules are sent by FedEx every two months and are taken daily without breaks. Participants and research assistants dealing with participants are blinded to the dose schedule. Data on adherence to the treatment protocol is monitored weekly using REDCap surveys. This treatment stage is the longest, lasting 8 months, with participants continuing to complete weekly outcome measures.

After eight months of study capsules, participants will enter a one-month endline phase where no medications are taken. Outcomes will still be completed once per week.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18 and 65
* Living in Alabama
* Meets ME-ICC criteria

Exclusion Criteria:

* Abnormal hepatic function
* Abnormal renal function
* Abnormal complete blood count
* Evidence of active or chronic systemic infection
* A1C > 9.0%
* Current opioid analgesic use
* Pregnant or plans to become pregnant during the study participation period
* Auto-immune disorder
* Enrolled in other experimental treatment study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
PROMIS Fatigue Short Form 7a | 10 months
  This will be measured using weekly surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Jarred Younger, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States